CLINICAL TRIAL: NCT00690924
Title: A Pilot Study of Oral Calcitriol in Patients at High Risk for Lung Cancer
Brief Title: Calcitriol in Preventing Lung Cancer in Smokers and Former Smokers at High Risk of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000596506; P30CA016056 (NIH); I 90206; NCT01896804 (obsolete NCT alias)
Record Dates: First submitted 2008-06-04; First posted 2008-06-05 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer; Precancerous Condition; Tobacco Use Disorder
Keywords: lung cancer; tobacco use disorder; squamous lung dysplasia
MeSH Terms: conditions — Lung Neoplasms; Precancerous Conditions; Tobacco Use Disorder | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Calcitriol (Experimental)
  Interventions: Drug: calcitriol; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: calcitriol — Oral
Other: laboratory biomarker analysis — Correlative Study
Other: pharmacological study — Correlative Study

SUMMARY:
RATIONALE: Calcitriol may prevent lung cancer in patients with metaplasia or dysplasia of the lungs.

PURPOSE: This clinical trial is studying the side effects and best dose of calcitriol in preventing lung cancer in current smokers and former smokers at high risk of lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the safety of calcitriol in patients at high risk of lung cancer.
* To determine the dose-limiting toxicities of calcitriol in these patients.

OUTLINE: Patients receive oral calcitriol on day 1. Courses repeat every 2 weeks for 3 months in absence of unacceptable toxicity.

Patients undergo blood collection periodically for pharmacokinetic and molecular analysis.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed squamous metaplasia or squamous dysplasia of the lungs by autofluorescence bronchoscopy within the past 5 years
* Must be a current or former smoker
* No evidence of concurrent disease with lung cancer or head and neck cancer

  * History of treated lung cancer or head and neck cancer treated with curative intent allowed, provided that there has been no evidence of disease for > 1 year

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Total granulocyte count > 1,500 x 10^9cells/L
* Platelet count > 100,000 x 10^9cells/L
* Calculated Creatinine clearance > 60 mL/min (using the Cockcroft-Gault formula)
* Calcium concentration 50-300 mg/24 hours
* Total bilirubin 0.2-1.3 mg%
* ALT/AST ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Albumin ≥ 2.5 g/dL
* Ionized serum calcium normal (1.19-1.29 mmol/L)
* Corrected serum calcium ≤ 10.2 mg/dL
* Willing to attend all scheduled study visits, complete all study questionnaires, and allow biological specimen collection, including a bronchoscopy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 1 month after completion of study therapy
* No life-threatening medical conditions that would preclude bronchoscopy, including but not limited to, any of the following:

  * Acute cardiac failure
  * Uncontrolled hypertension
  * Uncontrolled diabetes mellitus
  * Unstable coronary artery disease
* No severe metabolic disorders that would preclude calcitriol administration
* No history of any other malignancy within 3 years except for nonmelanoma skin cancer or cervical carcinoma in situ
* No history or evidence of kidney stones
* No patients who are susceptible to calcium-related dysrhythmias
* No known hypersensitivity to calcitriol
* No known allergies to tree nuts (i.e., almonds)

PRIOR CONCURRENT THERAPY:

* At least 2 months since prior and no concurrent calcium supplements
* Concurrent multivitamin supplement allowed provided the amount of vitamin D in the supplement is not in excess of the recommended daily dose
* No concurrent thiazides, phenobarbital, or digitalis
* No concurrent digoxin
* No concurrent bile acid binding drugs (i.e., cholestyramine, colestipol)
* No concurrent danazol or aluminum-based antacids
* No concurrent ketoconazole or other azole antifungals

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-07-17 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Reid, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcitriol
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Calcitriol
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Grade III-IV Toxicities or Any Grade II Toxicities Lasting More Than 2 Weeks
Description: Number of participants with Adverse Events, Grade II lasting more than two weeks or Grade III or higher, graded according to CTEP Version 4 of the NCI Common Terminology Criteria for Adverse Events (CTCAE) will be utilized for AE reporting.
  CTEP Version 4 of the CTCAE is identified and located at:
  http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm.
Time Frame: 3 months
Population: All treated and eligible patients
Measure: Number; unit: participants
Arm/Group | Calcitriol
Number analyzed (Participants) | 16
participants
  II | 1
  III | 0
  IV | 0
  V | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Calcitriol
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 13/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcitriol (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Eyelid irritation (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (5)
Constipation (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Calcium ionised increased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 7 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (5)
Headache (Nervous system disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT00690924/Prot_SAP_000.pdf